CLINICAL TRIAL: NCT05686694
Title: The Effect of Video Education Given on Pregnancy on Oral Glucose Tolerance Test Implementation Status, Knowledge, and Anxiety Level
Brief Title: Pregnancy on Oral Glucose Tolerance Test Implementation Status, Knowledge, and Anxiety Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Özlem D Bozkurt, PhD, Assoc. Prof., Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EGE-OZLEM-35; Gülcan KARABULUT (Other: Ege University, Women Health Nursing, master degree student)
Record Dates: First submitted 2022-12-21; First posted 2023-01-17 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-02

CONDITIONS: Gestational Diabetes
Keywords: Oral Glucose Tolerance Test; Primiparous Pregnant; Knowledge Level; Anxiety; Nursing
MeSH Terms: conditions — Diabetes, Gestational; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: single-blind, randomized controlled, experimental design
Who Masked: Participant
Masking Description: The research was planned as a single-blind randomized controlled experimental study. The homogeneity of the pregnant women in the education and control groups will be ensured according to age, education level and Instagram usage time. Considering the inclusion and exclusion criteria of the study, pregnant women will be divided into education and control groups by stratified randomization method. For this purpose, pregnant women who meet the criteria of the study will be assigned to the education and control group using a computer-assisted randomization program (https://www.random.org/). Pregnant women will not be informed about the groups they are in, and only the researcher will know which group they will be in, and single-blindness will be provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education Group (Experimental): 1. Follow-up (<24 weeks): "Questionnaire for Descriptive Characteristics of Pregnants" and "Informed Consent Form" and pretest application "Knowledge Level Form on the Pregnancy Diabetes and Oral Glucose Tolerance Test" will be made.
  2. Follow-up (<24. Week): Watching education videos:the education will end in 3 weeks. After that,post-test application "Knowledge Level Form on the Pregnancy Diabetes and Oral Glucose Tolerance Test" will be applied. They will be asked about their intention to have an OGTT.
  3. Follow-up (24-28. weeks): (Waiting after 75 mg dose is administered during OGTT): "State Anxiety Scale" will be applied. The OGTT implementation status of the pregnant woman will be recorded.
  4. Follow-up (30-34. weeks): 6 weeks after the video education, the "Knowledge Level Form on the Pregnancy Diabetes and Oral Glucose Tolerance Test" post-test application will be made.
  Interventions: Other: Video Education
- Control Group (No Intervention): 1. Follow-up (<24 weeks): "Questionnaire for the Introductory Characteristics of Pregnants" and "Informed Consent Form", and pre-test application "Knowledge Level Form on the Pregnancy Diabetes and Oral Glucose Tolerance Test" will be made.
  2. Follow-up (before OGTT implementation at 24-28 weeks): A posttest application will be made"Knowledge Level Form on Pregnancy Diabetes and Oral Glucose Tolerance Test". It will be asked about their intention to have an OGTT.
  3. Follow-up (24-28. weeks) (Waiting after 75 mg dose is administered during OGTT):"State Anxiety Scale" will be applied face-to-face while the pregnant woman is waiting after 75 mg dose is administered during the OGTT application while she is with the pregnant woman on the test day. In addition, the OGTT implementation status of the pregnant woman will be recorded.
  4. Follow-up (30-34 weeks): The post-test application of the "Knowledge Level Form on Pregnancy Diabetes and Oral Glucose Tolerance Test" will be made.

INTERVENTIONS:
Other: Video Education — Sharing of Planned Education Videos on Instagram In this research, the platform where planned video education will be shared was determined as "Instagram", which is the most used social media platform by pregnant women. In the Instagram user name "@ogttegitim" account, 6 education videos that will be created and shared.
  Arms: Education Group

SUMMARY:
This study was planned to examine the effect of video education on pregnancy for oral glucose tolerance test implementation status, knowledge and anxiety level. The research was planned as a single-blind randomized controlled experimental study.

DETAILED DESCRIPTION:
Hypothesis; H0: There is no difference between the OGTT knowledge level scores of primiparous pregnant women who received and did not receive video education.

H1: There is a difference between the OGTT knowledge level scores of primiparous pregnant women who received and did not receive video education.

H0: There is no difference between the status of having the OGTT, primiparous pregnant women who received and did not receive video education.

H1: There is a difference between the status of having the OGTT, primiparous pregnant women who received and did not receive video education.

H0: There is no difference between the mean scores of the State Anxiety Scale according to the video education status of the primiparous pregnant women who had OGTT.

H1: There is a difference between the mean scores of the State Anxiety Scale according to the video education status of the primiparous pregnant women who had OGTT.

H1: The anxiety level of pregnant women who had OGTT was lower than those who did not receive video education.

The research was planned as a single-blind randomized controlled experimental study. The homogeneity of the pregnant women in the education and control groups will be ensured according to age, education level and Instagram usage time. Considering the inclusion and exclusion criteria of the study, pregnant women will be divided into education and control groups by stratified randomization method. For this purpose, pregnant women who meet the criteria of the study will be assigned to the training and control group using a computer-assisted randomization program (https://www.random.org/). Pregnant women will not be informed about the groups they are in, and only the researcher will know which group they will be in, and single-blindness will be provided.

Dependent Variables The OGTT knowledge level of the pregnant women, their OGTT implementation status and the State Anxiety Inventory score average constitute the dependent variables of the study.

Independent variables The planned video OGTT training given to primiparous pregnant women constitutes the independent variable of the study.

Intermediate Variables Socio-demographic characteristics of pregnant women (age, occupation, marital status, family type, place of residence for the longest time, education level, income status, husband's occupation, husband's education level, husband's income), obstetric characteristics (gestational week, height, pregnancy Weight gained, family history of diabetes, history of miscarriage, presence of polycystic ovary syndrome), level of OGTT knowledge (the status of receiving information about OGTT, the people from whom they received information, the sufficient amount of information) constitute the intermediate variables of the research.

Informed Consent Form,Questionnaire for Descriptive Characteristics of Pregnants,Intention and Status of OGTT Questionnaire, Knowledge Level Form on Gestational Diabetes and Oral Glucose Tolerance Test (OGTT),State Anxiety Scale, Education Video Evaluation Form (for pilot group), Nickname card will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Reading and understanding Turkish
* literate
* over 18 years old
* under 35 years old
* primiparous pregnant
* before 24 weeks of pregnancy
* having a computer or phone and able to access the internet
* using Instagram
* voluntarily agreed to participate in the study

Exclusion Criteria:

* have a diagnosis of chronic diabetes mellitus (DM)
* have an ectopic pregnancy,
* want to leave the study voluntarily,
* in the education group but do not watch all the education videos
* have miscarriage or preterm birth
* pregnant women who do not fill in the all forms in study
* cannot be contacted during the research
* who decide to continue their doctor's checkups in another hospital

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 114 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Knowledge Level Form on the Pregnancy Diabetes and Oral Glucose Tolerance Test | before 24. pregnancy weeks and 30-34. pregnancy weeks
  Pregnant women will respond to each information sentence by choosing one of the options "True", "False", "I don't know". It is planned that the form will consist of 25 or 30 items. The state of knowing the items before and after the education will be evaluated with a percentage.
State Anxiety Scale | 24-28. pregnancy weeks
  During the evaluation, a score between 1 (or -1) and 4 (or -4) is given for each item according to the positive or negative feature of the item, and the constant 50 is added to the total score to be obtained. The highest score is 80 and the lowest score is 20. The higher the total anxiety score, the higher the anxiety level of the person completing the inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Demirel Bozkurt, Assoc. Prof., Principal Investigator — Ege University Nursing Faculty
Locations (1):
- Sağlık Bilimleri Üniversitesi Sarıyer Hamidiye Etfal Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We would like to publish it as an article. It has not yet been published in a journal.